CLINICAL TRIAL: NCT07285551
Title: Impact of Specific Physiotherapy and Whole-Body Vibration on Spinal Parameters in Patients With Adolescent Idiopathic Scoliosis
Brief Title: Physiotherapy and Whole-Body Vibration in Adolescent Idiopathic Scoliosis
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Gdansk University of Physical Education and Sport (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: AWFiS/2025_11_PE
Record Dates: First submitted 2025-11-17; First posted 2025-12-16 (Actual); Last update posted 2025-12-16 (Actual); Status verified 2025-12

CONDITIONS: Scoliosis Idiopathic Adolescent Treatment; Whole-body Vibration

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Rigo Concept group (Active Comparator): Physiotherapy/exercieses according to the Rigo Concept, 5 days, 3 hour per day
  Interventions: Procedure: Rigo Concept group
- Rigo Concept with whole-body vibration group (Experimental): Physiotherapy/exercises according to the Rigo Concept combined with whole-body vibration, 5 days, 3 hour per day, supplemented with 3 x 3 minutes of WBV, frequency 25 Hz, amplitude 2 mm
  Interventions: Procedure: Rigo Concept with whole-body vibration group

INTERVENTIONS:
Procedure: Rigo Concept group — 5-day physiotherapy based on the Rigo Concept. It has four general principles of correction such as three-dimensional stable postural correction, expansion technique, muscle activation, and integration. Intervention last for 3 hours per day.
  Arms: Rigo Concept group
Procedure: Rigo Concept with whole-body vibration group — The same like in the Rigo Concept groupa and additionally in standing position with two poles from Rigo Concept they will be exposed to WBV on a Galileo Med25 platform. WBV will administer in 3 x 3-minute sessions per day at a frequency of 25 Hz and an amplitude of 2 mm.
  Arms: Rigo Concept with whole-body vibration group

SUMMARY:
The aim of this study is to assess how physiotherapy based on the Rigo Concept, combined with WBV, affects sagittal spinal curvatures, the angle of trunk rotation (ATR), and trunk symmetry in girls with AIS.

Participants undergo a 5-day individualized physiotherapy program. The exercises follow the four general principles of the Rigo Concept: three-dimensional postural correction, expansion technique, muscle activation, and integration. Therapy is delivered for 3 hours per day, with three 15-minute breaks. Additionally, participants in the Rigo Concept with WBV group perform exercises in a standing position using two poles while exposed to WBV on a Galileo Med 35 platform (Novotec Medical GmbH, Pforzheim, Germany) at a frequency of 25 Hz, with a peak-to-peak displacement of 2 mm. Each session includes three 3-minute bouts of vibration, with 3-minute rests between them. During WBV, participants perform exercises according to the principles of the Rigo Concept.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of the adolescent idiopathic scoliosis
* Written consent of a medical doctor for participation
* Female

Exclusion Criteria:

* thrombosis
* body implants
* musculoskeletal inflammation
* arthropathy
* tendonitis
* hernia
* disc herniation
* recent fractures
* kidney stones
* recent scars
* surgery
* rheumatoid arthritis
* neuropathy
* epilepsy
* previous spinal surgery
* injuries in the spine during the past six months
* injuries in the lower limbs during the past six months
* pain in the spine during the past six months
* pain in the lower limbs during the past six months
* for group with WBV additionally discomfort or felt unwell during vibration exposure

Ages: 8 Years to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 50 (Estimated)
Dates: Start 2025-12 (Estimated); Primary Completion 2025-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Measurements of the sagittal curvature of the spine | Before the first physiotherapy session and three hours after the last physiotherapy session
  The examination of spinal curvatures (degrees) in the sagittal plane is conducted using a Baseline digital inclinometer (MVS in Motion, Belgium). Measurements are taken in a relaxed standing position. The assessment includes evaluation of thoracic kyphosis (upper and lower parts), lumbar lordosis, and sacral slope. The procedure is as follows: 1) Thoracic kyphosis - the inclinometer is zeroed at the thoracolumbar junction (Th12-L1), and the value is recorded at the cervicothoracic junction (C7-Th1); 2) Lumbar lordosis - the inclinometer is zeroed at the lumbosacral junction (L5-S1), and the value is recorded at the thoracolumbar junction (Th12-L1); 3) Sacral slope - the inclinometer is zeroed in the horizontal position, and the value is recorded at the lumbosacral junction (L5-S1).
Measurements of the trunk symmetry | Before the first physiotherapy session and three hours after the last physiotherapy session
  For postural alignment (centimeters), the physician positions a plumb line at the level of the occipital prominence. Measurements are performed using a rigid millimeter ruler and are rounded to the nearest 0 or 5 mm, assessing the distance from the plumb line to the gluteal cleft. For the assessment of scapular height asymmetry, the inferior angles of the scapulae are marked bilaterally. A rigid ruler is placed across these points, and a scoliometer is positioned on the ruler to record the angle of inclination (degrees). The distances from the inferior angles of the scapulae to the line of spinous processes are measured on both the left and right sides using a rigid ruler, and the differences (centimeters) are then calculated.
Measurements of the angle of trunk rotation | Before the first physiotherapy session and three hours after the last physiotherapy session
  The measurements of the angle of trunk rotation in the transverse plane are conducted using a Baseline scoliometer (MoVeS, Poland). The angle of trunk rotation is assessed during the Adams forward bend test. The participant stands in a relaxed upright position and is instructed to keep their hands together and slowly bend forward, aiming their hands toward the center of support. The examiner records the angle (degrees) and direction (left/right) of trunk rotation at the proximal and main thoracic spine, thoracolumbar region, lumbar spine, and at the level of the posterior superior iliac spine.

CONTACTS AND LOCATIONS:
Overall Officials: Paulina Ewertowska, Study Chair — Gdansk University of Physical Education and Sport
Locations (1):
- Korrektiv, Gdansk, Poland

IPD SHARING:
Plan to Share IPD: No